CLINICAL TRIAL: NCT01835561
Title: A Phase 1, Open-Label, Two-Part Study to Evaluate the Pharmacokinetics of Pomalidomide (CC-4047) in Hepatically Impaired Male Subjects
Brief Title: Study to Evaluate Pharmacokinetics of Pomalidomide in Hepatically Impaired Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CC-4047-CP-009
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Clinical Pharmacology, Healthy Volunteer Study
Keywords: Hepatic, Liver disease; Pharmacokinetic; Healthy
MeSH Terms: conditions — Liver Diseases | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: Severe liver disease and healthy volunteer match (Experimental): Subjects with severe liver disease (Group 2) and healthy volunteer subjects (Group 1) matched to the subjects with liver disease
  Interventions: Drug: Pomalidomide
- Part 2: Mild and moderate Liver disease (Experimental): Subjects with moderate (Group 3) and/or mild (Group 4) liver disease
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — Single oral dose of 4-mg capsule
  Other Names: POMALYST®
  Arms: Part 1: Severe liver disease and healthy volunteer match
Drug: Pomalidomide — 4-mg capsule
  Other Names: POMALYST®
  Arms: Part 2: Mild and moderate Liver disease

SUMMARY:
This study is for research purposes only and will not treat any disease or condition you may have. The study is an open label and single dose study; open label means that you, the study doctor and study staff will know which study drug you are taking.

The purpose of this research study is to compare drug levels in the body of people with liver disease to drug levels in healthy people with a normal liver. In addition, the safety of the study drug will be studied. Information about any side effects (discomfort or decline in health) that may happen will be collected. The study drug will be given by mouth to subjects with liver disease and to healthy subjects.

In the body, drugs are normally removed by the liver with a smaller amount being removed by the kidneys. When the liver is not working as well as it should, the body may not be able to remove drugs from the body quickly.

The information from this study will be used to decide if the drug is safe in subjects with liver disease or if a lower dose of the study drug would be safer.

DETAILED DESCRIPTION:
The study will be conducted at more than one clinical site (2-3 clinical research sites) and designed to assess the impact of severe liver disease or hepatic impairment (Part 1, Group 1) on the PK of pomalidomide following oral administration of a single dose of 4 mg pomalidomide (the study drug). The study drug, pomalidomide (POMALYST®), has been approved by the United States Food and Drug Administration (FDA) to treat patients with multiple myeloma (MM). Patients with MM have bone marrow that produces a large number of abnormal cells. Pomalidomide is only available by prescription.

Since participants in this study do not have MM, pomalidomide is considered experimental for the purposes of this research study. Throughout this form, pomalidomide will be referred to as "the study drug."

Participation in this study will be in either the healthy group or the group with liver disease. For the group with the liver disease,the liver disease will be graded by the study doctor as being "severe," "moderate," or "mild." This will be done by the study doctor depending on medical history, physical examination, laboratory tests, and certain previous results of liver scans or liver biopsy.

The amount of the study drug in blood will be measured at certain times to how well the drug is broken-down or removed from the body. Blood samples approximately 1 teaspoon (approximately 5-6 mL) will be collected 13 times the following times to measure study drug levels in your blood:

• Predose (just before dosing), and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, and 48 hours after dose pomalidomide morning dose on Day 1.

This study will have two parts:

Part 1 will evaluate the study drug in subjects with severe liver disease (Group and healthy volunteer subjects (Group 1) matched to the subjects with liver disease. Part 2 will evaluate the study drug in subjects with moderate (Group 3) and/ mild (Group 4) liver disease.

Study participation will be in one part only (either Part 1 or Part 2). Part be conducted after the data from Part 1 is analyzed and reviewed and the doctor and the sponsor determine that there is a need to conduct Part 2.

The purposes of this study are:

* To measure and compare the levels of pomalidomide in the blood of male subjects with severe liver disease and their matched healthy volunteer subjects after taking one 4-mg capsule of pomalidomide.
* To measure and compare the levels of pomalidomide in the blood of male subjects with moderate or mild liver disease after taking one 4-mg capsule of pomalidomide.
* To study the impact of liver disease on the safety of a single dose of pomalidomide in male subjects with liver disease.

Approximately 16 male subjects will be enrolled in Part 1 of the study (8 healthy subjects and 8 subjects with severe liver disease). Approximately 16 male subjects will be in Part 2 of the study (8 subjects with mild liver disease and subjects with moderate liver disease). If both parts of the study are completed, a total of about 32 male subjects will be enrolled. The total time a participant will be in the study is about 1 month (from screening visit to end of study).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Matched Healthy Subjects (Group 1):

  1. Must understand and voluntarily sign a written informed consent document (ICD) prior to any study-related procedures being performed.
  2. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
  3. Must be male subjects of any race between 18 to 70 years of age, inclusive, with a body mass index between 18 and 37 kg/m2 (inclusive).
  4. Subjects must be in good health (at screening and baseline [Day -1]) as determined by the investigator on the basis of medical history, physical examination, clinical laboratory safety test results, vital signs, and 12 lead ECG.
  5. Clinical laboratory safety tests must be within normal limits or acceptable to the investigator (at screening and baseline [Day -1]), and in particular:

     a. Creatinine less than or equal to 1.5x upper limit of normal (ULN)
  6. Must be afebrile, with supine (after the subject has rested for at least 5 minutes) systolic blood pressure: 90 to 140 mmHg, supine diastolic blood pressure: 60 to 90 mmHg, and pulse rate: 40 to 110 bpm.
  7. Must have a normal or clinically acceptable 12-lead ECG. Male subjects must have a QTcF value ≤ 430 msec.
  8. Subjects (with or without vasectomy) must practice true abstinence* or agree to use double barrier contraception (ie, latex condom or any non-latex condom not made out of natural [animal] membrane [eg, polyurethane]) and one other method (eg, spermicide) when engaging in sexual activity with woman of child-bearing potential during study conduct, and for 28 days after the last dose of study medication.

     * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
  9. Must agree to refrain from donating sperm, blood or plasma (other than for this study) while participating in this study and for at least 28 days after the last dose of study drug.
  10. Subjects who have not performed strenuous physical activity for at least 72 hours prior to the dose of study drug and agree to not engage in strenuous physical activity throughout the study and until study completion (follow-up safety telephone call).
  11. Will be counseled about pregnancy precautions and risks of fetal exposure and agree to comply with the conditions described in the counseling document.

Inclusion Criteria for All Hepatically Impaired Subjects (Groups 2, 3 and 4):

1. Must understand and voluntarily sign a written informed consent form (ICF) prior to any study-related procedures being performed.
2. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Male subjects of any race between 18 to 70 years of age, inclusive, with a body mass index between 18 and 37 kg/m2 (inclusive).
4. Subjects must have severe, moderate, or mild hepatic impairment or cirrhosis due to chronic hepatic diseases and/or prior alcohol abuse (Groups 2, 3 and 4, respectively).
5. Creatinine less than or equal to 1.5X ULN.
6. Subjects should be enrolled into the group corresponding to the Child-Pugh classification score that most accurately reflects the most severe hepatic disease classification within the past 6 months (based upon past medical history or physical examination observations). Adequate documentation should be provided to substantiate the Child-Pugh score assigned to each subject.

   1. For Group 2 (severe hepatic impairment), if biopsy, laparoscopy or ultrasound is not performed prior to screening, subjects can be included only if they have chronic liver disease and objective evidence of portal hypertension (ascites diagnosed by imaging or varices), with a Child-Pugh score ≥10 and ≤13.
   2. Subjects in Group 3 (moderate hepatic impairment) are required to have confirmation of the diagnosis of cirrhosis made by biopsy, laparoscopy or ultrasound with a Child-Pugh score of 7 to 9, inclusive.
   3. Subjects in Group 4 (mild hepatic impairment) are required to have confirmation of the diagnosis of cirrhosis made by biopsy laparoscopy or ultrasound with a Child- Pugh score of 5 to 6, inclusive.
7. Subjects may be treated with diuretics for ascites; however, subjects with severe ascites at time of enrollment may only be included at the discretion of the investigator with agreement of the Sponsor.
8. Subjects must not have history of hepatorenal syndrome or hemolysis.
9. Subjects (with or without vasectomy) must practice true abstinence* or agree to use double barrier contraception (ie, latex condom or any non-latex condom not made out of natural [animal] membrane [eg, polyurethane]) and one other method (eg, spermicide) when engaging in sexual activity with woman of child-bearing potential during study conduct, and for 28 days after the last dose of study medication.

   * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
10. Must agree to refrain from donating sperm, blood or plasma (other than for this study) while participating in this study and for at least 28 days after the last dose of study drug.
11. Will be counseled about pregnancy precautions and risks of fetal exposure and agree to comply with the conditions described in the counseling document .
12. Subjects are medically stable for at least 1 month before pomalidomide administration with clinically acceptable physical exam, clinical lab tests, vital signs, and 12-lead ECG consistent with the underlying stable mild, moderate or severe impaired liver condition as judged by the investigator.
13. Subjects must be free of acute major illness within one month prior to dosing or acute illness within 14 days prior to dosing, with the exception of hepatic impairment and related illnesses as judged by the investigator.
14. Subjects who have not performed strenuous physical activity for at least 72 hours prior to the dose of study drug and agree to not engage in strenuous physical activity throughout the study and until study completion (follow-up safety telephone call).

Exclusion Criteria:

* Exclusion Criteria for Matched Healthy Subject (Group 1)

  1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, known hypersensitivity to a member of the class of IMiDs, or other major disorders.
  2. Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
  3. Used any prescribed systemic or topical medication within 30 days of the first dose administration, unless Sponsor agreement is obtained.
  4. Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, unless Sponsor agreement is obtained.
  5. Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME), including but not limited to: bariatric procedure, irritable bowel syndrome (IBS), peptic ulcer(s),cholecystectomy, and chronic liver disease.
  6. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
  7. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual (DSM) within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs.
  8. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or positive alcohol screen.
  9. Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody, or have a positive result to the test for HIV antibodies at Screening.
  10. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
  11. Smokes more than 10 cigarettes, or consumes the equivalent in tobacco, per day.
  12. Subjects who are part of the staff personnel or family members of the investigational study staff.
  13. Subjects who, for any reason, are deemed by the investigator to be inappropriate for this study, including subjects who are unable to communicate or to cooperate with the investigator or the clinical staff.
* Exclusion Criteria for Hepatically Impaired Subject (Groups 2, 3 and 4)

  1. Any serious medical condition (excluding hepatic impairment and related complications), clinically significant laboratory abnormality not related to hepatic impairment and related complications, or psychiatric illness that would prevent the subject from signing the ICD and participating in the study.
  2. Any unstable clinically significant illness other than moderate or severe hepatic impairment within 3 months prior to the subject signing the ICD.
  3. Hepatic encephalopathy with time-disorientation, somnolent, stuporous, place disorientation, hyperactive reflexes, rigidity, slower electroencephalography (EEG) waves, unrousable coma, no personality/behavior, decerebrate, and slow 2-3 counts per second (cps) delta activity.
  4. Have a positive test result for Human Immunodeficiency Virus (HIV) antibodies.
  5. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
  6. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual (DSM) within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs.
  7. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
  8. Smokes more than 10 cigarettes, or consumes the equivalent in tobacco, per day.
  9. Subjects who are part of the staff personnel or family members of the investigational study staff.
  10. Subjects who, for any reason, are deemed by the investigator to be inappropriate for this study, including subjects who are unable to communicate or to cooperate with the investigator or the clinical staff.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-08-16 (Actual); Study Completion 2014-08-21 (Actual)

PRIMARY OUTCOMES:
C max | At predose (0-hour) and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, 40 and 48 hours post dose
  Observed maximum concentration; PK parameter for plasma pomalidomide
T max | At predose (0-hour) and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, 40 and 48 hours post dose
  Time to Cmax
Area Under the Curve Time Zero to time(AUC0-t) | At predose (0-hour) and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, 40 and 48 hours post dose
  Area under the plasma concentration-time curve from time zero to time t, where t is the last measurable time point
Area Under the Curve (AUCinf) ; from time 0 to infinity | At predose (0-hour) and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, 40 and 48 hours post dose
  Area under the plasma concentration-time curve from time zero extrapolated to infinity; PK parameter for plasma pomalidomide
t ½: Terminal Half Life | At predose (0-hour) and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, 40 and 48 hours post dose
  Estimate of the terminal elimination half-life in plasma 5. delay between time of administration and absorption
CL/F: apparent clearance | At predose (0-hour) and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, 40 and 48 hours post dose
  Apparent total plasma or serum clearance of drug after oral administration
Vz/F: apparent volume of distribution | At predose (0-hour) and at 0.25, 1, 2, 2.5, 4, 6, 8, 12, 24, 30, 40 and 48 hours post dose
  Apparent volume of distribution during terminal phase after oral / extravascular administration

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs). | 1 month (from screening visit to end of study follow-up telephone call).
  An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values (as specified by the criteria below), regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene Corporation
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota